CLINICAL TRIAL: NCT02082665
Title: An Open-label Phase 1 Study to Evaluate the Effects of Dabrafenib (GSK2118436) on the Single Dose Pharmacokinetics of an OATP1B1/1B3 Substrate and of a CYP3A4 Substrate in Subjects With BRAF V600 Mutation Positive Tumors
Brief Title: Effects of Dabrafenib on the Single Dose Pharmacokinetics (PK) of Rosuvastatin and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200919
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Cancer
Keywords: rosuvastatin; BRAF V600; Melanoma; dabrafenib; midazolam
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — Midazolam; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): On Day 1 subjects will simultaneously receive single dose of Rosuvastatin 10 mg tablet and Midazolam 3 mg syrup administered orally in the morning.
  Interventions: Drug: Rosuvastatin10 mg tablet; Drug: Midazolam 3 mg syrup; Drug: Dabrafenib 75 mg capsule

INTERVENTIONS:
Drug: Rosuvastatin10 mg tablet — Commercially available Rosuvastatin 10 mg tablets will be supplied. Single oral dose of Rosuvastatin 10 mg will be administered on Day 1, 8 and 22
Drug: Midazolam 3 mg syrup — Commercially available Midazolam syrup will be supplied.Single oral dose of Midazolam 3 mg syrup will be administered on Days 1, 8 and 22
Drug: Dabrafenib 75 mg capsule — Dabrafenib 75mg will be supplied in the form of capsules. Oral dose Dabrafenib 150 mg (2 x 75 mg) BID will be administered at 12 h apart on Days 8 through 22 and 150 mg (2 x 75 mg) OD on Day 23.

SUMMARY:
This is an open-label, multi-center, fixed sequence study in subjects with BRAF V600 mutation positive tumors. Subjects will receive single oral doses of 10 milligram (mg) of rosuvastatin and 3 mg of midazolam in the morning of Day 1 (alone), Day 8 (with first dose of dabrafenib 150 mg), and Day 22 (during repeat dose dabrafenib 150 mg twice daily [BID]). Dabrafenib 150 mg BID will be administered from Day 8 to Day 23. Blood samples for PK analysis will be obtained over 32 hours post-dose on Day 1, Day 8, and Day 22. The last dose of dabrafenib will be taken in the morning of Day 23 and the last blood sample in the evening of Day 23. Subjects will be considered to have completed the study once the 32 hour PK sample has been collected on Day 23. Once they have completed the study, eligible subjects may have the option to enter study BRF114144, an open-label roll-over study of dabrafenib (no follow-up visit required) and continue receiving dabrafenib.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent.
* BRAF V600 mutation-positive tumor: as confirmed by a Clinical Laboratory Improvement Amendments (CLIA) approved local laboratory or equivalent.
* Male or female between 18 to 65 years of age, inclusive, at the time of signing the informed consent form;
* Capable of compliance with the requirements and restrictions listed in the consent form;
* Body weight >= 45 kilogram (kg) and a body mass index >= 19 kilogram per squaremeter (kg/m^2)and <40 kg/m^2 (inclusive);
* Able to swallow and retain orally administered medication
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1. NOTE: Subjects with a performance status of 2 can be enrolled if the subject's confinement to bed and inability to carry out work activities is due solely to cancer-related pain, as assessed by the Investigator.
* Adequate baseline organ function defined as: absolute neutrophil count >= 1.2 x 10^9/Liter (L); hemoglobin>=9 gram per deciliter (g/dL); platelets >= 75 x 10^9/L; prothrombin time /international normalized ratio and partial thromboplastin time =<1.3 x ULN; serum bilirubin=<1.5 times upper limit of normal (ULN); aspartate aminotransferase and alanine aminotransferase =<2.5 times ULN; serum creatinine=<1.5 mg/dL or calculate creatinine clearance >= 50 milliliter per minute; Left ventricular ejection fraction>= lower limit of normal by echocardiography.
* Women of child-bearing potential must be willing to practice acceptable methods of birth control. Additionally, women of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study medication.

Exclusion Criteria:

* History of another malignancy with exceptions below, or any malignancy with confirmed activating RAS mutation. Exception: (a) Subjects who have been successfully treated and are disease-free for 5 years, (b) a history of completely resected non-melanoma skin cancer, (c) successfully treated in situ carcinoma, (d) chronic lymphocytic leukemia in stable remission, or (e) indolent prostate cancer (definition: clinical stage T1 or T2a, Gleason score <=6, and prostate-specific antigen <10 nanogram per milliliter) requiring no or only anti-hormonal therapy, are eligible. Note: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility.
* Cancer therapy (chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) or investigational anti-cancer drugs within the last 3 weeks, or chemotherapy without delayed toxicity within the last 2 weeks, preceding the first dose of study medication.
* Unresolved clinically significant toxicity greater than Grade 2 from previous anti-cancer therapy
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Current use of therapeutic warfarin. NOTE: Low molecular weight heparin and prophylactic low-dose warfarin are permitted
* Any prohibited medication(s) or herbal preparation as described in the protocol or requires any of these medications during the study.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to dabrafenib, rosuvastatin, and midazolam, or excipients that contraindicate their participation; or have an allergy to cherries.
* Pregnant or nursing females.
* A history or evidence of cardiovascular risk including any of the following:
* A QT interval corrected for heart rate using the Bazett's formula (QTcB) >=480 millisecond (msec);
* A history or evidence of current clinically significant uncontrolled arrhythmias;
* A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
* A history or evidence of current >=Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines
* Abnormal cardiac valve morphology (>=grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
* Patients with intra-cardiac defibrillators
* Presence of active GI disease or other condition (e.g., small bowel or large bowel resection) that will interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, contact the GSK Medical Monitor.
* Subjects with COPD or subjects with increased risk of respiratory depression
* Subjects with narrow angle glaucoma
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus, or Hepatitis C Virus infection.
* Subjects with brain metastases are excluded if their brain metastases are: Symptomatic; Treated (surgery, radiation therapy) but not clinically and radiographically stable one month after local therapy, OR; Asymptomatic and untreated but > 1 cm in the longest dimension. Subjects with small (<= 1 cm in the longest dimension), asymptomatic brain metastases that do not need immediate local therapy can be enrolled. Subjects on a stable dose of corticosteroids for more than one month, or those who have been off corticosteroids for at least 2 weeks can be enrolled. Subjects must also be off of enzyme-inducing anticonvulsants for more than 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02-19; Primary Completion 2016-07-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of rosuvastatin and midazolam | Day 1, Day 8 (initiation of dabrafenib dosing) and Day 22 (steady state)
  Blood samples will be collected for assessment of PK parameters including maximum observed concentration (Cmax), time to Cmax (tmax), and area under the concentration-time curve from pre-dose extrapolated to infinite time (AUC[0-infinity])

SECONDARY OUTCOMES:
Secondary PK parameters of rosuvastatin and midazolam | Day 1, Day 8 (initiation of dabrafenib dosing) and Day 22 (steady state)
  Blood samples will be collected for assessment of PK parameters including area under the concentration-time curve to time of last measurable concentration (AUC[0-t]), area under the concentration-time curve from time zero to a time point determined from the data (AUC (partial), terminal phase half-life (t1/2)
PK parameters of dabrafenib and dabrafenib metabolites | Day 8 and 22; pre-dose, 1 hour (hr), 2 hr, 8 hr and 24 hr after dose
  Blood samples will be collected for assessment of concentration of dabrafenib and its metabolites
Number of subjects with adverse events as a measure of safety and tolerability | Screening and up to 10 days post last dose. Skin exams may continue through 6 months post study.
  AE is defined as Any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Changes in clinical laboratory measurements to access safety | Screening, Day 1, Day 22 and Follow-up
  Any abnormal laboratory test results (haematology, clinical chemistry, or urinalysis)
Changes in vital sign measurements to access safety | Screening, Day 1, Day 2, Day 8, Day 9, Day 22 , Day 23 and Follow-up
  Vital sign measurements will include systolic and diastolic blood pressure, respiratory rate, pulse rate and pulse oximetry Vital signs should be measured after sitting in a semi-supine position for at least 5 min.
Change from baseline in cardiac assessments | Screening, Day 1, Day 22,and Follow-up
  Cardiac assessments include 12-lead Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Lebanon, New Hampshire, United States
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville

REFERENCES:
- [Derived] Nebot N, Won CS, Moreno V, Munoz-Couselo E, Lee DY, Gasal E, Bouillaud E. Evaluation of the Effects of Repeat-Dose Dabrafenib on the Single-Dose Pharmacokinetics of Rosuvastatin (OATP1B1/1B3 Substrate) and Midazolam (CYP3A4 Substrate). Clin Pharmacol Drug Dev. 2021 Sep;10(9):1054-1063. doi: 10.1002/cpdd.937. Epub 2021 May 1. PMID 33932130